CLINICAL TRIAL: NCT06480474
Title: Internet-based Treatment for Depression: a Randomized Controlled Trial Comparing Therapist Support and Peer-support Using an Online Forum.
Brief Title: Internet-based Treatment for Depression
Acronym: IBAT-D
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Fribourg (Other)
Collaborators: University of Bern (Other); Indian Institute of Technology (Unknown); Gaia AG (Industry); Haute école d'Ingénierie et d'Architecture de Fribourg (Unknown)
Responsible Party: Principal Investigator, Chantal Martin Soelch, Prof. Dr., University of Fribourg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-D0112
Record Dates: First submitted 2024-06-17; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Depression
Keywords: depression; online intervention; internet-based treatment; online study; peer-support; randomized control trial; India; Switzerland
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: We will use a controlled randomized design with 3 conditions (1. Online program, 2. Online program and online forum, 3. Wait list). Participants will be assessed at 4 time points: before the beginning of the intervention (T0, baseline), at 4 weeks mid-treatment (T1), after the intervention, at 8 weeks (T2), and at the follow-up, that is 3 months post-intervention (T3).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental): The first experimental group will have access to an online self-help program for depression. The program Deprexis® is a self-help, web-based intervention that proposed various modules to face depression. They will have access to the program for 8 weeks. They are asked to complete the modules as many times as they wish and to use to program at least 30 minutes, 1 or 2 times a week. They will be assessed at baseline (T0), mid-intervention (4-weeks, T1), post-intervention (8-weeks, T2) and for the follow-up (3 months post intervention, T3). They will be asked to complete online questionnaires.
  Interventions: Device: Deprexis
- Second Experimental group (Active Comparator): The second experimental group will have access to both the online program as well as an online forum in which they will be divided into a group of 10 and they will be requested to ask, respond, and share their experiences with other participants. They will have access to the program and to the online forum for 8 weeks. They are asked to complete the modules as many times as they wish and to use to program at least 30 minutes, 1 or 2 times a week. They will be assessed at baseline (T0), mid-intervention (4-weeks, T1), post-intervention (8-weeks, T2) and for the follow-up (3 months post intervention, T3). They will be asked to complete online questionnaires.
  Interventions: Device: Deprexis; Device: Deprexis with online forum
- Control group (No Intervention): The control intervention is a wait list control group that will, after the 8 weeks of treatment, have access to the online self-help program and will complete questionnaires (the same as the two experimental groups), reward task at baseline, at 8-weeks and at the follow-up (3 months post-intervention).

INTERVENTIONS:
Device: Deprexis — The internet-based self-help program used in this study, Deprexis, contains 10 modules ( based on different psychotherapeutic approaches, consistent with a cognitive-behavioral perspective) and accessible at any time via regular internet browsers on laptops, computers, tablets, or smartphones through a secure website. Participants can repeat all modules as often as they wish after completing the full sequence once.
  Arms: Experimental group; Second Experimental group
Device: Deprexis with online forum — Those in this group will have access to deprexis ( same as the first group) as well as an online forum built for the study. This forum will feature a general discussion page where participants can ask and answer questions, and they will be divided into groups of 10 to share experiences if they wish. Additionally, there will be subforums related to specific modules of the program. Participants can share their experiences and ask questions related to the modules. A moderator will regularly check to ensure no personal or sensitive information is disclosed and will ask questions weekly to encourage contributions to the forum.
  Arms: Second Experimental group

SUMMARY:
The overall aim of the present project is to test the efficacy of a validated Internet-based self-help program for depression developed in Germany in the French part of Switzerland. The program has shown to be efficacious in different trials with major depression and depression as a comorbidity of another disorder (e.g., gambling addiction, epilepsy). The objectives of this project are:

Primary Objective: To test the effects of the self-help web-based program on depressive symptoms in French-speaking individuals in Switzerland.

Secondary Objective A: To test the effects of the online program on reward responses for individuals with depressive symptoms.

Secondary Objectives B and C: To test the effects of the role of peer-to-peer support using an online forum in addition to an online program (B) and comparison between Switzerland and India (C).

This project can inform clinicians about what they can offer as a treatment to individuals, either in combination with psychotherapy or when there is no quick or direct access to a psychotherapist. The study promises to have a direct practical significance for people suffering from depression.

DETAILED DESCRIPTION:
Depression is one of the most frequent mental disorders that affect society and individuals psychologically and financially. The text revision of the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5-TR) defines characterized depression as a minimum of 2 weeks of low mood or loss of interest in daily activities, accompanied by vegetative, motor, and cognitive symptoms. Depressed individuals may also have suicidal thoughts or tendencies. However, not everyone receives adequate care and there is a treatment gap. The causes of the treatment gap are diverse and include the difficulty in accessing treatment, the lack of mental health specialists in a region or a country, the fear of stigmatization, cultural beliefs about mental health, etc.. Technologies such as Internet-based self-help interventions are promising to reduce the burden of depression and to address the treatment gap. Several meta-analyses found that these interventions are effective in reducing depression. Internet-based self-help interventions are easily available, can be utilized regardless of time and location, and can be provided to a large population simultaneously. Although Switzerland has a well-developed mental health care, the treatment gap for depression in Switzerland is estimated to be 51% and depression represents a strong societal burden. The main aim of this study will be to examine the efficacy of a web-based self-help intervention for depression in the French-speaking part of Switzerland, in a randomized clinical trial.

Moreover, anhedonia is a core symptom of depression. It is defined as a loss of pleasure or a lack of reactivity when faced with pleasurable stimuli . Hedonic capacity decreases with depression, such as a reduced reactivity to pleasant cues or diminished reward responsiveness . Reward processes are shown to induce positive or pleasurable experiences . Specifically, there might be a strong association between the presence of anhedonia in depressed patients and dysfunction of the reward system . One secondary objective (A) of this project is to examine reward responses and sensitivity in individuals with depressive symptoms and more specifically, the effect of an online intervention for depression on reward responses. Finally, whereas the effect of therapist support (in the form of guidance during the treatment) in internet-based self-help programs is well investigated, the role of peer support within internet-based self-help has not yet been fully understood. There is evidence suggesting that patients' mutual exchange via integrated discussion forums can increase the efficacy of Internet-based treatments and could help to overcome adherence issues of Internet-based self-help programs. Further secondary objectives (B and C) of this study are to investigate the effects of the role of peer-to-peer support using an online forum in addition to an online program and comparison between Switzerland and India.

ELIGIBILITY:
Inclusion Criteria:

* Read and signed inform consent.
* Older than 18 years old
* Have access to a computer or laptop or tablet with an internet connection.
* Sufficient French language skills
* Fulfil the criteria of characterised depression according to the M.I.N.I diagnostic interview.
* Provide emergency contact before intervention.

Exclusion Criteria:

* Active suicidal plans (score higher on the suicide item or report suicidal plan in the diagnostic interview)
* Have a history of psychotic disorder or bipolar disorder.
* Have changed their dosage of prescribed medication for anxiety or depression in the last month before the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | Post-Intervention (+8 weeks +/- 2 weeks)
  The primary outcome measures are symptoms of depression at post-treatment, that is after 8 weeks. Depressive symptoms will be measured with the Patient Health Questionnaire (PHQ-9) to assess the symptoms of depression.

SECONDARY OUTCOMES:
Secondary Objective A | Baseline (0 week) , Mid-intervention (+4 weeks +/- 2 weeks), Post-Intervention (+8 weeks +/- 2 weeks), Follow-up (+20 weeks +/- 2 weeks)
  The secondary objective A aims to test the effects of the online program on reward responses for individuals with depressive symptoms. We will assess constructs at Baseline (T0), mid-intervention (4 weeks, T1), post-intervention (8 weeks, T2), and follow-up (3 months after intervention, T3). We will also use a reward task described below. Outcomes associated with the reward task will be evaluated, including anhedonia and reward sensitivity.
  Fribourg Reward Task: This task measures reaction times, accuracy, and mood reactions to both monetary and social rewards.
  Snaith-Hamilton Pleasure Scale (SHAPS): This scale measures the ability to experience pleasure, covering four areas of hedonic experience: interest/pastimes, social interaction, sensory experience, and food/drink.
  Behavioral Inhibition System/Behavioral Activation System (BIS/BAS): This self-reported questionnaire measures activation and inhibition systems, or sensitivity to punishment and reward.
Secondary Objective B and C | Baseline (0 week), Post-Intervention (+8 weeks +/- 2 weeks)
  The secondary objectives B and C aim to test the effect of the role of peer-to-peer support with an online forum in addition to an online program (B) and in comparison, between Switzerland and India (C). For this objective, we will assess perceived social support at Baseline (T0) and at post-treatment (T2). This will be evaluated by using:
  Perceived Social Support (PSS). The PSS is a self-report questionnaire, which assesses the perception of support from family, friends, and a significant other.
Additional/Exploratory Outcomes | Post-Intervention (+8 weeks +/- 2 weeks), Follow-up (+20 weeks +/- 2 weeks)
  We aim to study treatment effects on comorbid depression symptoms, focusing on anxiety assessed via the Generalized Anxiety Disorder Scale (GAD) for symptoms like nervousness, worry, trouble relaxing, restlessness, irritability, and fear. Additionally, we'll explore how positive outcomes such as self-efficacy (GSES), quality of life (SF-12), and self-esteem (RSE) positively impact depression symptoms. We'll also investigate the influence of stress, trauma, and pain using the Perceived Stress Scale-Short Version (PSS), Somatic Symptom Scale (SSS-8), PTSD Checklist for DSM-5 (PCL-5), and Childhood Trauma Questionnaire-Short Form (CTQ-SF). Lastly, we'll evaluate client satisfaction, usability, and working alliance using the System Usability Scale (SUS) for user experience and satisfaction, and the Client Satisfaction Questionnaire (CSQ) for service satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Chantal Martin Soelch, Fribourg, Switzerland

REFERENCES:
- [Background] Kessler RC, Wang PS. The descriptive epidemiology of commonly occurring mental disorders in the United States. Annu Rev Public Health. 2008;29:115-29. doi: 10.1146/annurev.publhealth.29.020907.090847. PMID 18348707
- [Background] Tandon T, Piccolo M, Ledermann K, Gupta R, Morina N, Martin-Soelch C. Relationship between behavioral and mood responses to monetary rewards in a sample of Indian students with and without reported pain. Sci Rep. 2022 Nov 24;12(1):20242. doi: 10.1038/s41598-022-24821-2. PMID 36424426
- [Background] Tanner JA, Davies PE, Overall CC, Grima D, Nam J, Dechairo BM. Cost-effectiveness of combinatorial pharmacogenomic testing for depression from the Canadian public payer perspective. Pharmacogenomics. 2020 Jun;21(8):521-531. doi: 10.2217/pgs-2020-0012. Epub 2020 Apr 17. PMID 32301648
- [Background] Pizzagalli DA, Iosifescu D, Hallett LA, Ratner KG, Fava M. Reduced hedonic capacity in major depressive disorder: evidence from a probabilistic reward task. J Psychiatr Res. 2008 Nov;43(1):76-87. doi: 10.1016/j.jpsychires.2008.03.001. Epub 2008 Apr 22. PMID 18433774
- [Background] Rojas LM, Bahamon M, Wagstaff R, Ferre I, Perrino T, Estrada Y, St George SM, Pantin H, Prado G. Evidence-based prevention programs targeting youth mental and behavioral health in primary care: A systematic review. Prev Med. 2019 Mar;120:85-99. doi: 10.1016/j.ypmed.2018.12.009. Epub 2019 Jan 2. PMID 30610888
- [Background] Snaith RP, Hamilton M, Morley S, Humayan A, Hargreaves D, Trigwell P. A scale for the assessment of hedonic tone the Snaith-Hamilton Pleasure Scale. Br J Psychiatry. 1995 Jul;167(1):99-103. doi: 10.1192/bjp.167.1.99. PMID 7551619
- [Background] Andersson G, Cuijpers P. Internet-based and other computerized psychological treatments for adult depression: a meta-analysis. Cogn Behav Ther. 2009;38(4):196-205. doi: 10.1080/16506070903318960. PMID 20183695
- [Background] Berger T, Hammerli K, Gubser N, Andersson G, Caspar F. Internet-based treatment of depression: a randomized controlled trial comparing guided with unguided self-help. Cogn Behav Ther. 2011;40(4):251-66. doi: 10.1080/16506073.2011.616531. PMID 22060248
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Cuijpers P, Cristea IA, Karyotaki E, Reijnders M, Hollon SD. Component studies of psychological treatments of adult depression: A systematic review and meta-analysis. Psychother Res. 2019 Jan;29(1):15-29. doi: 10.1080/10503307.2017.1395922. Epub 2017 Nov 7. PMID 29115185
- [Background] Karyotaki E, Efthimiou O, Miguel C, Bermpohl FMG, Furukawa TA, Cuijpers P; Individual Patient Data Meta-Analyses for Depression (IPDMA-DE) Collaboration; Riper H, Patel V, Mira A, Gemmil AW, Yeung AS, Lange A, Williams AD, Mackinnon A, Geraedts A, van Straten A, Meyer B, Bjorkelund C, Knaevelsrud C, Beevers CG, Botella C, Strunk DR, Mohr DC, Ebert DD, Kessler D, Richards D, Littlewood E, Forsell E, Feng F, Wang F, Andersson G, Hadjistavropoulos H, Christensen H, Ezawa ID, Choi I, Rosso IM, Klein JP, Shumake J, Garcia-Campayo J, Milgrom J, Smith J, Montero-Marin J, Newby JM, Breton-Lopez J, Schneider J, Vernmark K, Bucker L, Sheeber LB, Warmerdam L, Farrer L, Heinrich M, Huibers MJH, Kivi M, Kraepelien M, Forand NR, Pugh N, Lindefors N, Lintvedt O, Zagorscak P, Carlbring P, Phillips R, Johansson R, Kessler RC, Brabyn S, Perini S, Rauch SL, Gilbody S, Moritz S, Berger T, Pop V, Kaldo V, Spek V, Forsell Y. Internet-Based Cognitive Behavioral Therapy for Depression: A Systematic Review and Individual Patient Data Network Meta-analysis. JAMA Psychiatry. 2021 Apr 1;78(4):361-371. doi: 10.1001/jamapsychiatry.2020.4364. PMID 33471111
- [Background] Klein JP, Barthel B, Berger T, Moritz S. Feasibility, effectiveness and safety of the self-management intervention deprexis in routine medical care: Results of an uncontrolled observational study. Internet Interv. 2020 Dec;22:100341. doi: 10.1016/j.invent.2020.100341. Epub 2020 Aug 27. PMID 32874927
- [Background] Meyer B, Berger T, Caspar F, Beevers CG, Andersson G, Weiss M. Effectiveness of a novel integrative online treatment for depression (Deprexis): randomized controlled trial. J Med Internet Res. 2009 May 11;11(2):e15. doi: 10.2196/jmir.1151. PMID 19632969
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Derived] Tandon T, Berger T, Meyer B, Khaled OA, Gupta R, Martin-Soelch C. Exploring cross-cultural effectiveness of internet-based depression treatment (IBAT-D) with peer-to-peer support vs. without across WEIRD and non-WEIRD samples: a research protocol for a randomized controlled trial. Trials. 2025 Dec 11;26(1):569. doi: 10.1186/s13063-025-09377-6. PMID 41382119